CLINICAL TRIAL: NCT01529216
Title: An Advanced Configuration (The Third Generation) of the DIAMOND System for the Treatment of T2DM Patients - A Randomized, Double Blind Study
Brief Title: Efficacy Study of the DIAMOND System to Treat Type 2 Diabetes Mellitus
Acronym: RUBY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaCure Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MC CP TAN2011- 014
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DIAMOND System; T2DM; Randomized study; Electrical stimulation; Fundus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrical signal ON (Experimental): Subjects randomized to this group (Group A) will receive electrical stimulation delivered to the fundus for 24 months.
  Interventions: Device: DIAMOND System
- Sham (Sham Comparator): Subjects randomized to this group (Group B) will have their device in "turned off" mode for the first 12 months (48 weeks) after implant. Then the device will be turned ON and these subjects will receive therapy for the remaining 12 months of the study.
  Interventions: Device: DIAMOND System

INTERVENTIONS:
Device: DIAMOND System — Electrical stimulation to the fundus

SUMMARY:
The study purpose is to demonstrate the benefit of a simplified version of the DIAMOND System (A third Generation) in comparison to a sham treatment in terms of Glycemic control, measured as A1c, FBG and Post-Prandial Glucose levels.

The study hypothesis is that HbA1c will show greater improvement in patients receiving 12 months of therapy by the DIAMOMD System than in patients not receiving this therapy.

DETAILED DESCRIPTION:
The study protocol will also apply measures to better understand the mechanism of action of the effect.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 21 through 70 years of age
* Body mass index ≥28 and ≤ 45 (kg/m2)
* Type 2 diabetes duration more than 6 months and less than 10 years.
* A baseline measurement (visit BL1) of HbA1c between ≥ 7.5% and ≤ 10.5%,
* Type 2 diabetic subjects treated for at least 3 months with one or more maximum tolerable dosage of anti-diabetic agent (Any of the following: Sulfonylurea, Metformin, thiazolinedione (TZD), DPP-4 inhibitors).
* Stable anti-hypertensive and lipid-lowering medication for at least one month prior to enrollment, if taken
* Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods
* Ability and willingness to perform required study and data collection procedures and adhere to operating requirements of the System
* Alert, mentally competent, and able to understand and willing to comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial
* Able to provide voluntary informed consent

Exclusion Criteria:

* Injectable anti-diabetic therapy within the last 3 months (such as insulin and/or GLP-1 receptor agonists)
* Taking medications known to affect gastric motility such as narcotics (chronic use) and anticholinergics/antispasmodics
* Any gastric or upper GI surgery
* Experiencing severe and progressing diabetic complications (i.e. retinopathy not stabilized, nephropathy with macroalbuminuria)
* Prior wound healing problems
* Diagnosed with past or current psychiatric condition that may impair his or her ability to comply with the study procedures
* Use of anti-psychotic medications
* Diagnosed with an eating disorder such as bulimia or binge eating
* Obesity due to an endocrinopathy (e.g. Cushing disease, Hypothyroidism not treated)
* Hiatal hernia requiring surgical repair or a paraesophageal hernia
* Pregnant or lactating
* Diagnosed with impaired liver function (liver enzymes 3 times greater than normal)
* Any prior bariatric surgery
* Any history of pancreatitis
* Any history of peptic ulcer disease within 10 years of enrollment
* Diagnosed with Gastroparesis or other GI motility disorder
* Use of active medical devices (either implantable or external) such as ICD, pacemaker, drug infusion device, or neurostimulator (either implanted or worn). Subjects using an external active device who are able and willing to avoid use of the device during the study may be enrolled.
* Cardiac history that physician /surgeon feels should exclude the subject from the study.
* Use of another investigational device or agent in the 30 days prior to enrollment
* A history of life-threatening disease within 5 years of enrollment
* Any additional condition(s) that in the Investigator"s opinion would warrant exclusion from the study or prevent the subject from completing the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 months
  The primary end point will be the difference, at 12 months, in HbA1c change from baseline, between the pts treated with the active signal compared to patients treated with a Sham System.

SECONDARY OUTCOMES:
HbA1c | 6 months
  The difference, at 6 months in HbA1c change from baseline, between the pts treated with the active signal compared to patients treated with a Sham System.
GI hormones (C-peptide, Glucagon, Ghrelin, GLP-1, PYY, Gastrin and Somatostatin) | 6 and 12 months
  To detect differences in the pattern of meal-related release of GI hormones (slope / area under the curve, etc)between the treatment and the control groups, as analyzed by repeated-measures ANOVA. Glucose, insulin and the following GI hormones will be measured prior and post meal consumption: C-peptide, Glucagon, Ghrelin, GLP-1, PYY, Gastrin and Somatostatin.
Metabolic parameters (fasting and post Prandial glucose, blood pressure, lipids and cholesterol, weight and waist circumference) | 6 and 12 months
  The difference in metabolic parameters at 6 and 12 months from baseline between the two arms. Including: fasting and post Prandial glucose, blood pressure, lipids and cholesterol, weight and waist circumference.
Triglycerides | Baseline
  The effect of the TG level at baseline on treatment efficacy
HbA1c | 24 months
  The change in HbA1c from baseline to 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan W.M. Greve, MD, Principal Investigator — Atrium medisch centrum METC, Heerlen, The Netherlands; Chevallier, MD, Principal Investigator — Hôpital GEORGES POMPIDOU 20 Rue Leblanc 75015 Paris, France
Locations (2):
- Hospital Georges Pompidou, Paris, France
- Atrium Medisch Centrum, Heerlen, Netherlands

REFERENCES:
- See also: MetaCure — http://www.metacure.com